CLINICAL TRIAL: NCT03702699
Title: Detecting Auricular Points Among Patients With Knee Osteoarthritis by A Novel Auricular Point Detector (APD): A Pilot Diagnostic Accuracy Study
Brief Title: Detecting Auricular Points in KOA by a Novel APD
Acronym: APD-KOA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); City University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: SCM-ACU-01
Record Dates: First submitted 2018-10-03; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis, Knee
Keywords: auricular point detection; knee osteoarthritis; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- KOA group: Patients in this group will receive auricular point detection which is accomplished by the novel auricular point detector device. There is no addition to the patient's routine care.
  Interventions: Device: Auricular point detector
- Control group: This group includes healthy subject, for whom no treatment will be performed. Only auricular point detection by the auricular point detector will be conducted.
  Interventions: Device: Auricular point detector

INTERVENTIONS:
Device: Auricular point detector — This device is only for auricular detection. No additional intervention will be delivered.

SUMMARY:
This is a pilot diagnostic accuracy study conducted to assess the diagnostic ability of a novel APD for auricular point detection among patients with knee osteoarthritis (KOA), as compared with an already commercialized device.

DETAILED DESCRIPTION:
The present study is a pilot diagnostic accuracy study conducted to assess the diagnostic ability of a novel APD for auricular point detection among patients with knee osteoarthritis, as compared with an already commercialized device. The investigators will test if the novel APD could provide a more reliable and quantifiable diagnosis than traditional devices currently available in the market; They will also use the APD device to test whether the cutaneous electrical impedance detected from the corresponding auricular points by the novel device is the lowest in the knee and lower limb area in the KOA population. As a pilot study, 12 patients with KOA will be recruited from the Department of Anesthesiology, Queen Mary Hospital, the University of Hong Kong. 12 healthy subjects will be recruited from the university community. Auricular acupoint detection will be accomplished with the new device and a control device. The electrical impedance will be measured and recorded. Patient's condition will also be evaluated by the Knee Injury and Osteoarthritis Outcome Score (KOOS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The specificity and sensitivity of the auricular point detection by the APD device will be calculated. Cohen's kappa coefficient (κ) will be used to test the inter-methods reliability, test-retest reliability, and inter-tester reliability. Moreover, the Pearson Correlation Coefficient will be used to test the correlation between the electrical impedance of the auricular point of knee and the KOOS score and WOMAC score.

ELIGIBILITY:
Inclusion Criteria:

* Average daily knee pain >=5 point measured by a 10-point VAS scale;
* Diagnosed KOA of any reason;
* The different patient categories;
* Patients with knee osteoarthritis enrolled for knee arthroplasty, osteotomies around the knee, cartilage repair, or anterior cruciate ligament-deficient knees enrolled for anterior cruciate ligament reconstruction;
* Surgical plan in the coming month after inclusion;
* Provide written inform consent;
* Free of any other diagnosed psychological conditions;

Exclusion Criteria:

* with any other diseases such as cardiovascular, renal, neurological, digestive, hepatic, respiratory disease;
* Pregnancy or lactation;
* Participation in a clinical study that may interfere with participation in this study;
* History of or current tobacco, alcohol use;
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study;
* Unable to provide written informed consent due to any reason;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: KOA patients with surgical schedule will be referred to this study by an anesthesiologist from the inpatient or outpatient unit of the Department of Anesthesiology Queen Mary Hospital.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
cohen's kappa coefficient | baseline
  The Cohen's kappa coefficient is a statistical test used to validate the inter-method reliability, test-retest reliability and inter-observer reliability of the device.

SECONDARY OUTCOMES:
the Visual Analogue Scale (VAS) | baseline
  The VAS is a common instrument used to measure pain intensity. The scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates worst pain possible.
the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a 24-item instrument used to measure pain and joint function among patients with osteoarthritis. For each item, there is a Likert 5-point scale (ranging from 0 to 4), where 0 = none and 4 = extremely. It includes three major domains, including pain, stiffness, and physical function. The total score is calculated as the sum of the items chosen divided by 96.
the Knee Injury and Osteoarthritis Outcome Score (KOOS) | baseline
  Knee Injury and Osteoarthritis Outcome Score (KOOS) is a validated 42-item global knee score suitable for comparison of patients with knee complaints attributable to different causes. A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
self-developed questionnaire on patient's attitude towards complementary therapies for pain management | baseline
  This is a self-developed questionnaire which includes 10 items aiming to survey patient's attitude towards the use of complementary therapies for pain management. This questionnaire only includes descriptive answers to be choose. The percentage for each choice will calculated.
The diagnostic specificity of the device | baseline
  The specificity test is a test to validate the ability of a diagnosis to tell the 'non-disease' among those without the disease.
The diagnostic sensitivity of the device | baseline
  The sensitivity test is a test to validate the ability of a diagnosis to tell the 'disease' among those with the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lixing Lao, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, HKU, Hong Kong, INTL, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing depends on the discretion of participants and principal investigator.